CLINICAL TRIAL: NCT03141047
Title: Lifespan Integration After Sexual Trauma, a Randomized Treatment Study
Brief Title: Lifespan Integration After Sexual Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insamlingsstiftelsen Wonsa, World of No Sexual Abuse (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1001
Record Dates: First submitted 2016-03-25; First posted 2017-05-04 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Symptoms of Post Traumatic Stress Disorder (PTSD)
Keywords: Sexual trauma, Lifespan Integration
MeSH Terms: conditions — Sexual Trauma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifespan Integration (Experimental): This arm is given one session of Lifespan Integration. Differences on Impact of Event Scale from the first measurement at inclusion and the second measurement 20 +/- 3 days after the first measurement, and after treatment, is analyzed and compared with the results from the Group on waiting list. A third measurement and comparison is being made 6 months +/- 6 weeks after the first measurement at inclusion.
  Interventions: Other: Lifespan Integration
- Waiting list (No Intervention): This arm gets no treatment, and differences on Impact of Event Scale from the first measurement at inclusion at the second measurement 20 +/- 3 days after, without treatment, is analyzed and compared with the results from the treatment Group. A third measurement and comparison is being made 6 months +/- 6 week after the first measurement at inclusion.

INTERVENTIONS:
Other: Lifespan Integration — A protocol based psychological treatment method
  Arms: Lifespan Integration

SUMMARY:
A new psychological trauma treatment method is tested on a population (n 100) of adult women who have been sexually traumatized at one specific time 0-5 years before they enter the study.

DETAILED DESCRIPTION:
One treatment session is given with the psychological treatment method Lifespan Integration (LI). The main outcome is change on Impact of Event Scale (IES) before and after the treatment. The change is analyzed and compared with the change on Impact of Event Scale (IES) among the people on the waiting list arm. Self-rating questionnaires are being used 5+/-3 days before treatment, 20 +/-3 days after treatment, and 6 months +/- 6 weeks after the first measurement.

ELIGIBILITY:
Inclusion Criteria:

* Sexual trauma 1-5 years before inclusion
* understanding Swedish, read and spoken

Exclusion Criteria:

* Psychotic symptoms
* drug abuse
* neuropsychiatric diagnoses ADHD and asperger

Ages: 15 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Change of Points on Impact of event scale before and after Lifespan Integration treatment after a sexual trauma | 3 weeks
  One treatment is given, and change is measured 20 +/- 3 days after treatment.

SECONDARY OUTCOMES:
Change of Points of GHQ12 | 3 weeks
  General Health Questionnaire 12
Change of Points of Stressful Events Survey PTSD Short Scale (NSESS) | 3 weeks
  Questionnaire
Self Rated Health and Sickness Questionnaire | 3 weeks
  10 items on current symptoms of sickness

OTHER OUTCOMES:
Change of Points on Impact of event scale before and after Lifespan Integration treatment | 6 months
  One treatment is given, and change is measured two weeks after treatment and six months after treatment.
Change of Points of Stressful Events Survey PTSD Short Scale (NSESS) | 6 months
  Questionnaire
Self Rated Health and Sickness Questionnaire | 6 months
  10 items on current symptoms of sickness

CONTACTS AND LOCATIONS:
Overall Officials: Axel C Carlsson, Docent, Principal Investigator — Karolinska Institutet
Locations (1):
- World of no sexual abuse, Wonsa, Stockholm, Stortorget 3, Sweden

REFERENCES:
- [Derived] Rajan G, Wachtler C, Lee S, Wandell P, Philips B, Wahlstrom L, Svedin CG, Carlsson AC. A One-Session Treatment of PTSD After Single Sexual Assault Trauma. A Pilot Study of the WONSA MLI Project: A Randomized Controlled Trial. J Interpers Violence. 2022 May;37(9-10):NP6582-NP6603. doi: 10.1177/0886260520965973. Epub 2020 Oct 21. PMID 33084475